CLINICAL TRIAL: NCT00530933
Title: Prospective Randomised Placebo Controlled Study Into Percutaneous and Transcutaneous Tibial Nerve Stimulation for Faecal Incontinence
Brief Title: Tibial Nerve Stimulation for Faecal Incontinence
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: London North West Healthcare NHS Trust (Other)
Collaborators: Uroplasty, Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 07/Q0405/13
Record Dates: First submitted 2007-09-15; First posted 2007-09-18 (Estimated); Last update posted 2007-09-18 (Estimated); Status verified 2007-09

CONDITIONS: Fecal Incontinence
MeSH Terms: conditions — Fecal Incontinence

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Sham Comparator): Sham tibial nerve stimulation
  Interventions: Procedure: Sham transcutaneous tibial nerve stimulation
- 2 (Experimental): Percutaneous tibial nerve stimulation
  Interventions: Procedure: Percutaneous posterior tibial nerve stimulation
- 3 (Experimental): Transcutaneous tibial nerve stimulation
  Interventions: Procedure: Transcutaneous tibial nerve stimulation

INTERVENTIONS:
Procedure: Percutaneous posterior tibial nerve stimulation — Once weekly for 30 minutes
  Arms: 2
Procedure: Transcutaneous tibial nerve stimulation — 30 minutes once weekly
  Arms: 3
Procedure: Sham transcutaneous tibial nerve stimulation — Once weekly for 30 minutes
  Arms: 1

SUMMARY:
The purpose of this study is to determine whether tibial nerve stimulation is an effective treatment for faecal incontinence.

DETAILED DESCRIPTION:
Faecal incontinence is a common problem, affecting approximately 2% of the adult general population. Initial management involves dietary advice, anti-diarrhoeal medication, and behavioural therapy. In those who have not benefited from these conservative techniques sacral nerve stimulation is an established and effective treatment for faecal incontinence. This treatment involves using electrical pulses to stimulate the S3 nerve root - a nerve at the bottom of the back. These are the nerves which supply the lower end of the bowel, and the anal sphincter. It is believed that it is stimulation of the sensory fibres heading back towards the spinal cord at this level which is important for the therapeutic effect. To stimulate the sacral nerves however requires two operations under general anaesthetic, and surgical implantation of an expensive nerve stimulator.

The tibial nerve also contains fibres that arise from the S3 part of the spinal cord. Electrical stimulation of the tibial nerve will therefore send sensory information back to the same region of the spinal cord as sacral nerve stimulation. The tibial nerve is much more easily accessible on the inside of the ankle, and this allows stimulation to be carried out as an outpatient and without the need for surgery. It can be performed either percutaneously (with a fine needle placed through the skin to sit next to the nerve), or transcutaneously.

Tibial nerve stimulation has been successfully used for patients with urinary incontinence. There are small studies looking at tibial nerve stimulation for faecal incontinence which both show a benefit, but these studies are not controlled. We aim to determine in a randomised controlled trial whether either percutaneous or transcutaneous tibial nerve stimulation is an effective treatment for faecal incontinence.

ELIGIBILITY:
Inclusion Criteria:

* Over 18
* Incontinence to solid or liquid faeces

Exclusion Criteria:

* Previous congenital or acquired spinal injury, spinal tumour or spinal surgery
* Neurological diseases, such as diabetic neuropathy, multiple sclerosis and Parkinson's disease
* Peripheral vascular disease
* Diabetes mellitus
* Congenital anorectal malformations
* Previous rectal surgery (rectopexy / resection) done < 12 months ago (24 months for cancer)
* Present evidence of external full thickness rectal prolapse
* Chronic bowel diseases such as inflammatory bowel disease
* Chronic diarrhoea, uncontrolled by drugs or diet
* Anatomical limitations that would prevent successful placement of an electrode
* Previous use of transcutaneous electrical nerve stimulation Stoma in situ

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2007-09; Study Completion 2009-04 (Estimated)

PRIMARY OUTCOMES:
The difference in the percentage of patients with a 20% reduction in episodes of faecal incontinence between the placebo and treatment groups. | 14 weeks

SECONDARY OUTCOMES:
The difference in the improvements in the St Mark's incontinence score, quality of life scales, and physiological parameters between the treatment and placebo groups. | 14 weeks
The difference in the improvements in the urinary symptoms between placebo and treatment groups. | 14 weeks

CONTACTS AND LOCATIONS:
Overall Officials: James Hollingshead, MRCS, Principal Investigator — London North West Healthcare NHS Trust; Carolynne Vaizey, MD FRCS FCS, Study Director — London North West Healthcare NHS Trust
Locations (1):
- St Mark's Hospital, London, United Kingdom

REFERENCES:
- [Derived] George AT, Kalmar K, Sala S, Kopanakis K, Panarese A, Dudding TC, Hollingshead JR, Nicholls RJ, Vaizey CJ. Randomized controlled trial of percutaneous versus transcutaneous posterior tibial nerve stimulation in faecal incontinence. Br J Surg. 2013 Feb;100(3):330-8. doi: 10.1002/bjs.9000. PMID 23300071